CLINICAL TRIAL: NCT03603873
Title: Preoperative Anxiety Level, Premeds and General Anaesthetic Proceedings
Brief Title: Preoperative Anxiety Level, Premedications and General Anaesthetic Proceedings
Status: Completed | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: PZ17011
Record Dates: First submitted 2018-07-19; First posted 2018-07-27 (Actual); Last update posted 2018-07-27 (Actual); Status verified 2018-07

CONDITIONS: Anxiety; Premedication; General Anaesthetic
Keywords: Anxiety; Premedication; general anaesthetic
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients

SUMMARY:
Although it seems obvious that the high level of preoperative anxiety may affect intraoperative anaesthetic requirements and recovery adversely, there are several contradictory studies about this subject. Furthermore, the effects of anxiolytic premedication are actually disputed: sedative premedication is widely administered but little clinical evidence supports its use.

We want to evaluate the effects of pre-procedure anxiety for propofol needs in patients receiving general anaesthetic procedure. We also want to know if premedication is useful according to the preoperative anxiety level, in order to determine if a sub-group of patients benefit from it.

DETAILED DESCRIPTION:
This study will be carried out in solely at the institute of CHU de Reims, France (Reims Teaching Hospital) from March 2017 to May 2017. Selected patients will be over the age of 18, among those receiving general anaesthesia for surgery. Demographic data and medical history will be collected after written consent. Before the anaesthetic procedure, an APAIS questionnaire (Anxiety evaluation form) will be filled out by each patient.

The medical, anaesthetic and surgical care will not be changed. In the operating room, we will proceed with anaesthetic induction following a medical protocol according to the practice of our hospital (TCI Target Controlled Infusion or manual induction): the propofol infusion or injection is started with an initial effect-site concentration or dose and increased step by step until patients present the clinical en points defined as LOC (loss of consciousness, i.e. no response to a verbal command).

The effect-site concentration of propofol, induction time required for a loss of consciousness (LOC), and preoperative incidents will be recorded by an anaesthetist student nurse and will be recorded in a data book.

After surgery, we will record any secondary effect attributable to premedication.

The day after surgery, patients will be assessed with the EVAN-G questionnaire. Statistical analysis will be done in sub-groups with variance analysis. We will also do multivariate regression analysis according to the type of premedication, demographic data, preoperative variable and preoperative anxiety level. If the number of included patients allows it, we will do propensity score matching for premedication.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years old
* surgery with general anaesthetic, programmed, in emergency or ambulatory
* Cognitive level adequate to submit APAIS - EVANG form
* General anaesthetic induction procedure using propofol

Exclusion Criteria:

* ASA 4 level
* Patient refusal
* pregnancy
* Rapid Sequence Induction (ISR)
* General Anaesthetic induction procedure using another drug than propofol (thiopental - etomidate)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with scheduled or urgent surgical procedure
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Actual)
Dates: Start 2017-03-03 (Actual); Primary Completion 2017-05-24 (Actual); Study Completion 2017-05-24 (Actual)

PRIMARY OUTCOMES:
Preoperative anxiety level | Day 0
  this outcome will be interpreted according to the preoperative anxiety level (APAIS score)
Premeds | Day 0
  this outcome will be interpreted according to the use or not of premeds

CONTACTS AND LOCATIONS:
Locations (1):
- Damien JOLLY, Reims, France